CLINICAL TRIAL: NCT02870426
Title: Collection and Characterisation of Human Olfactory Ensheathing Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 16.0069
Record Dates: First submitted 2016-04-26; First posted 2016-08-17 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-03

CONDITIONS: Spinal Cord Injury
Keywords: Olfactory ensheathing cells
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Cells and tissue from olfactory ensheathing cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1A:: Donors after brainstem death (DBDs) undergoing solid organ donation
  Interventions: Procedure: Frontal Craniotomy and retrieval of OBs
- Group 1B:: Donors after brainstem death (DBDs) considered unsuitable for solid organ donation
  Interventions: Procedure: Frontal Craniotomy and retrieval of OBs
- Group 2:: Neurosurgical patients undergoing anterior cranial surgery in which the olfactory nerve (ON) is cut as part of the surgical procedure. The OB of the concomitant severed ON would be donated.
  Interventions: Procedure: OB Retrieval During Anterior Cranial Surgery

INTERVENTIONS:
Procedure: Frontal Craniotomy and retrieval of OBs — For Group 1A the craniotomy will occur during organ retrieval for transplantation under aseptic technique. For Group 1B it would occur as a separate surgical procedure prior to palliation under full asepsis.
  Groups: Group 1A:; Group 1B:
Procedure: OB Retrieval During Anterior Cranial Surgery — Group 2: The patients routine anterior cranial surgery would proceed as planned without change to the surgical procedure. In the event that the ON had to be sacrificed for the purposes of surgery the OB of the concomitant nerve would be retrieved.
  Groups: Group 2:

SUMMARY:
We aim to retrieve olfactory bulbs (OBs) from suitable human donors. We have defined two groups who will qualify:

Group 1 - Deceased Donors:

1A: Donors after brainstem death (DBDs) undergoing solid organ donation

1B: Donors after brainstem death (DBDs) considered unsuitable for solid organ donation

Group 2 - Living Donors:

Neurosurgical patients undergoing anterior cranial surgery in which the olfactory nerve (ON) is cut as part of the surgical procedure. The OB of the concomitant severed ON would be donated.

We aim to optimise OB collection and Olfactory Ensheathing Cell (OEC) culture and storage. We will study the effects of patient diagnosis, age, cause of death (if applicable), co-morbidities and warm ischaemic time on cell survival and regenerative function.

In future studies we aim to store OECs in a GMP facility and transplant OECs into patients with spinal cord injuries.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a devastating condition. To date there is no treatment to improve outcome. There is limited regenerative capacity of the central nervous system (CNS), such that damaged neurons and severed axons are not replaced.

A substantial body of evidence suggests that olfactory ensheathing cells (OECs) obtained from olfactory bulbs (OBs) facilitate neuronal regeneration in rodents and humans with SCI. Indeed, transplanting autologous OECs from an OB into the injury site improved neurological outcome in a patient with SCI.

Harvesting autologous OBs to culture OECs has several disadvantages:

1. If the OECs do not grow in vitro, the transplantation is abandoned;
2. The retrieval procedure exposes a paralysed patient to the risks of craniotomy;
3. Excising an OB can impair the sense of smell; and
4. The number of OECs obtained is limited to one OB.

Investigators will collect human OECs from suitable donors which we have defined as two groups. Group 1 patients will be brain dead donors identified by the neuro-intensive care team as potential candidates for solid organ donation. The OBs will be retrieved as near to death as possible. Group 2 patients will be living donors undergoing elective neurosurgery in which the olfactory nerve is sacrificed as part of that procedure.

There are two OBs located at the anterior skull base, responsible for transmitting the sensation of smell from the nose to the brain. Obtaining OECs requires a craniotomy (opening the skull) to remove the OBs.

PHASE 1 will be divided into 2 stages. In stage 1 we will culture OECs and characterise them in the central laboratory. We aim to determine how the yield of OECs and their regenerative properties are affected by freeze-thaw, time left at room temperature and time left at 40C before culture as well as patient age. Each harvested sample will be transferred to the lab for further processing. Processing includes but is not limited to histological fixation, sectioning and staining, cell culture and storage. Some OECs will be frozen in liquid nitrogen to determine whether they can indeed be stored. In stage 2 we will transfer OECs outside St. George's to a GMP facility (to be determined). In the GMP facility, the OECs will be processed and stored according to the optimised conditions we have determined.

In PHASE 2, the OECs will be transplanted into patients with SCI.

ELIGIBILITY:
Inclusion criteria:

Group 1 - Deceased Donors 1A

1. Diagnosis of brainstem death, AND
2. Consent from next of kin (NoK) for organ donation
3. Consent from NoK for removal of olfactory bulbs (OBs)
4. Coroner's consent for removal of OBs (when needed).

1B

1. Diagnosis of brainstem death, AND
2. Contraindications for solid organ donation
3. Consent from NoK for removal of OBs
4. Coroners consent for removal of OBs (when needed)

Group 2 - Living Donors

1. Patients having anterior cranial surgery in which the ON may be cut or removed as part of the procedure.
2. Consent from the operating surgeon to remove the OB of the corresponding ON in the event it is cut during the operation
3. Consent from the patient for removal of the OB of the corresponding ON in the event it is cut during the operation

Exclusion criteria:

1. Children (<18 years old)
2. Damage to anterior skull base including OBs
3. Meningitis

And applicable to group 2 only:

Patients unable to consent for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Deceased brain dead donors and living patients undergoing anterior cranial surgery in which the ON may be sacrificed as routine part of the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Ability to culture olfactory ensheathing cells from human donors | 10-15 days
  Number of olfactory ensheathing cells cultured per olfactory bulb at days 10-15 in vitro.

SECONDARY OUTCOMES:
Effect of cause of death for Group 1 donors | 10-15 days
  Plot of cause of death vs. Number of olfactory ensheathing cells cultured per olfactory bulb at days 10-15 in vitro.
Effect of patient age | 10-15 days
  Plot of patient age vs. Number of olfactory ensheathing cells cultured per olfactory bulb at days 10-15 in vitro.
Effect of freeze/thaw cycles | 10-15 days
  Plot of number of freeze/thaw cycles vs. Number of olfactory ensheathing cells cultured at days 10-15 in vitro.
Effect of storage in liquid nitrogen | up to 1 month
  Plot of Number of olfactory ensheathing cells cultured at days 10-15 in vitro when cells are cultured fresh vs. after one week and one month storage in liquid nitrogen.
Effect of time from extraction to culture at room temperature | 1 month
  Plot of time from extraction to culture vs. Number of olfactory ensheathing cells cultured.
Effect of time from extraction to culture at 4 deg C | 1 month
  Plot of time from extraction to culture at 4 deg C vs. Number of olfactory ensheathing cells cultured.

CONTACTS AND LOCATIONS:
Overall Officials: Marios Papadopoulos, FRCS (SN), Principal Investigator — St George's, University of London; Samira Saadoun, PhD, Principal Investigator — St George's, University of London
Locations (1):
- St George's Hospital, London, Tooting, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tabakow P, Jarmundowicz W, Czapiga B, Fortuna W, Miedzybrodzki R, Czyz M, Huber J, Szarek D, Okurowski S, Szewczyk P, Gorski A, Raisman G. Transplantation of autologous olfactory ensheathing cells in complete human spinal cord injury. Cell Transplant. 2013;22(9):1591-612. doi: 10.3727/096368912X663532. PMID 24007776
- [Result] Miedzybrodzki R, Tabakow P, Fortuna W, Czapiga B, Jarmundowicz W. The olfactory bulb and olfactory mucosa obtained from human cadaver donors as a source of olfactory ensheathing cells. Glia. 2006 Nov 1;54(6):557-65. doi: 10.1002/glia.20395. PMID 16917854
- [Result] Raisman G. Olfactory ensheathing cells and repair of brain and spinal cord injuries. Cloning Stem Cells. 2004;6(4):364-8. doi: 10.1089/clo.2004.6.364. PMID 15671664
- [Result] Li Y, Decherchi P, Raisman G. Transplantation of olfactory ensheathing cells into spinal cord lesions restores breathing and climbing. J Neurosci. 2003 Feb 1;23(3):727-31. doi: 10.1523/JNEUROSCI.23-03-00727.2003. PMID 12574399
- [Result] Keyvan-Fouladi N, Li Y, Raisman G. How do transplanted olfactory ensheathing cells restore function? Brain Res Brain Res Rev. 2002 Oct;40(1-3):325-7. doi: 10.1016/s0165-0173(02)00215-1. PMID 12589931
- [Result] Raisman G. Olfactory ensheathing cells - another miracle cure for spinal cord injury? Nat Rev Neurosci. 2001 May;2(5):369-75. doi: 10.1038/35072576. PMID 11331921
- Available data/document: Individual Participant Data Set — http://www.stgeorges.nhs.uk — The project documents will be available directly from the research team. Please e-mail Dr Florence Hogg fhogg@sgul.ac.uk